CLINICAL TRIAL: NCT01564173
Title: Characterization of LV Hemodynamics During Epicardial and Endocardial Pacing
Brief Title: Dependence of LV Hemodynamics on Pacing Site
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 644
Record Dates: First submitted 2012-03-24; First posted 2012-03-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- VT Ablation: Patients undergoing epicardial mapping and ablation procedure for a ventricular tachycardia

SUMMARY:
The purpose of this study is to evaluate the effects of epicardial and endocardial pacing at each side of the left ventricular (LV) segments on cardiac hemodynamics in patients with impaired LV function undergoing epicardial ablation and mapping procedure. Hemodynamic function will be assessed during a pacing protocol with a pressure catheter inserted in the LV.

ELIGIBILITY:
Inclusion Criteria:

* Patient is already indicated for epicardial mapping and ablation of arrhythmia(s) utilizing a transcutaneous subxiphoid approach
* Be in sinus rhythm
* Have LVEF < 40%
* Have the ability to provide informed consent for study participation and be willing and able to comply with the CIP (Clinical Investigational Plan) described evaluations

Exclusion Criteria:

* Have permanent AF
* Have pericardial disease
* Have a recent myocardial infarction within 40 days prior to enrollment
* Have undergone cardiac surgery or coronary revascularization procedure within 3 months prior to enrollment or be scheduled for such procedures
* Have had a recent CVA or TIA within 3 months prior to enrollment
* Be less than 18 years of age
* Be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for epicardial mapping and ablation of arrhythmia(s) utilizing a transcutaneous subxiphoid approach
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Invasive Dp/dt Max | Acute E.P. Procedure
  Variation on invasive Dp/dt max during dedicated pacing site

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Jais, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU, Bordeaux, France